CLINICAL TRIAL: NCT02589327
Title: Effects of Exercise on Cardiac Fat in Women With Obesity: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 504792C
Record Dates: First submitted 2015-10-14; First posted 2015-10-28 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2015-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise Intervention (Experimental): Hight intensity resistance training group
  Interventions: Other: Exercise Intervention
- Control (No Intervention): No-exercise control group

INTERVENTIONS:
Other: Exercise Intervention — The intervention will consist of 3 weeks of whole body circuit training (resistance training) where participants in the intervention group will perform 7 different exercises. The circuit will consist of 10 repetitions per exercise of 7 exercises: leg press, bent-over row, bench press, squats, dumbbell jump squats with raises, dead-lifts and weighted abdominal crunches, with approximately 30 sec of rest in between each exercise (based on the estimated time needed to move from one position to the next). Each participant will move through the circuit 3 times, with 2 to 3 minutes of rest between each round. Intensity will be 6-7 of RPE at the first set, and 9-10 at the third set.
  Arms: Exercise Intervention

SUMMARY:
Excessive cardiac fat accumulation have been recognized to be associate to increased cardiac and metabolic risk. The aim of this study the effects of exercise in cardiac fat content, cardiac function, physical fitness, and metabolic activity in obesity.

DETAILED DESCRIPTION:
Excessive cardiac fat accumulation have been recognized to be associate to increased cardiac and metabolic risk. More effective treatments are needed to induce changes in cardiac fat content, body composition, and cardiac fat metabolic activity that result in a reduction in cardiovascular risk in overweight and obese population. Despite this need, little is known about which mode, frequency, and duration of exercise will allow for greater reductions in cardiac fat, improvements in body composition, restoration of a healthy cardiac fat metabolic activity, and improvement on cardiovascular risk markers. The aim of this study the effects of exercise in cardiac fat content, cardiac function, physical fitness, and metabolic activity in obesity.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30-39.99
* White/Caucasian

Exclusion Criteria:

* Known health problems such as cardiovascular, pulmonary or metabolic disease will be excluded.
* Pregnant females.
* Any adults found taking medications that affect endocrine or cardiovascular function will also be excluded from the study.
* Participants that exercise more than three times per week or strength train more than twice per week.
* Individuals that have poor venous access or have expressed a fear of needles or having blood taken will also be excluded.
* Cigarette smoking (current or those who quit within the previous 6 months
* Hypertension
* Diabetics
* MRI exclusion criteria must be observed: must complete a safety checklist that is designed to identify metal in your body that could pose a hazard during scanning. Some forms of metal are acceptable (e.g., dental fillings after 1970). Tattoos are generally not exclusionary, unless they have been inked with metallic dyes. All metal must be removed from your body. All female subjects, prior to scanning, are required to complete a pregnancy test. Must NOT be claustrophobic or have a history of claustrophobia

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Changes in Cardiac fat volumes | 2 assessment points: at baseline and week 4
  Cardiac fat volumes will be assessed by means of Magnetic Resonance Imaging

SECONDARY OUTCOMES:
Changes in Vascular function | 2 assessment points: at baseline and week 4
  Vascular function will be assessed by means of Arterial Tonometry
Changes in Cardiorespiratory Function | 2 assessment points: at baseline and week 4
  Cardiorespiratory Function will be assessed on a treadmill test with a 12-lead EKG. Protocol: Modified Bruce (A baseline stage will be added)
Changes in Muscular Strength | 2 assessment points: at baseline and week 4
  Muscular Strength in upper and lower extremities will be assessed by 1 repetition maximum (1RM) test on Bench Press and Leg Press
Changes in Body Composition | 2 assessment points: at baseline and week 4
  Body Composition will be assessed using Dual-energy x-ray absorptiometry
Changes in Diet | 5 assessment points: baseline, week 1, 2, 3, and 4
  Diet will be assessed using the ASA24h recall (http://epi.grants.cancer.gov/asa24/)
Changes in Spontaneous Physical Activity | Baseline and week 4
  Spontaneous Physical Activity will be assessed using accelerometers Actical.
Changes in Oxidative stress markers | 5 assessment points: pre-post during session 1, pre-post during session 9, and pre week 4.
  Blood will be collected and processed in order to assess oxidative stress markers

CONTACTS AND LOCATIONS:
Overall Officials: Maria Fernandez del Valle, PhD, Principal Investigator — Texas Tech University
Locations (1):
- Kinesiology and Sport Management, Lubbock, Texas, United States